CLINICAL TRIAL: NCT00683891
Title: FazaClo Outcomes in the Control of Schizophrenia (FOCUS)
Brief Title: FazaClo Outcomes in the Control of Schizophrenia (FOCUS) Study Survey
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: Azur Pharma, Inc (Industry)
Other Study IDs: FOCUS
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Weight Gain; Sialorrhea
Keywords: FOCUS; Weight gain; Sialorrhea; Treatment refractory schizophrenia; FazaClo; Treatment resistant schizophrenia; clozapine; Hypersalivation
MeSH Terms: conditions — Weight Gain; Sialorrhea; Schizophrenia, Treatment-Resistant | interventions — Clozapine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: FazaClo (clozapine, USP) ODT

SUMMARY:
AZUR Pharma has received several reports from practicing psychiatrists prescribing FazaClo showing that FazaClo patients start losing body weight instead of keep gaining it, after being switched from other clozapine products or other atypical antipsychotics treatments. Another important clinical observation reported by doctors is a considerable reduction in hypersalivation when FazaClo administration is compared to other antipsychotic treatments. Based on the findings described above, and on the real need for effective and safer treatments for schizophrenia, AZUR Pharma has decided to design and conduct an observational study in a large number of patients taking FazaClo to prove the received clinical reports from physicians. Better understanding and evaluation of these beneficial findings are necessary to provide physicians information for improved treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* Patients with treatment-resistant schizophrenia currently being treated with Clozaril or generic clozapine for at least 3 months
* Patients with treatment-resistant schizophrenia who failed to respond adequately to treatment with at least 2 courses of standard drug treatments for schizophrenia, either because of insufficient effectiveness or the inability to achieve an effective dose due to intolerable adverse effects from those drugs
* Males and females of 18 years of age or older
* Females of childbearing potential using a reliable form of contraception
* Ability to comply with the required WBC/ANC monitoring schedule
* Ability to follow physician's instructions
* Signed informed consent by patient or legal guardian

Exclusion Criteria:

* Phenylketonurics
* Females of childbearing potential not using a reliable form of contraception
* Women who are pregnant or want to become pregnant
* Nursing
* Patients allergic to clozapine or any othe ingredient contained in FazaClo tablets
* Patients who have previously experienced a severe adverse reaction to clozapine
* Patients previously excluded from taking clozapine due to a higher risk of developing white blood cell disorders
* Clinical significant medical condition that the physician believes may increase the patient's risk of participating int he study (e.g., severe cardiac disorder, epilepsy)
* Concomitant medications that may be contraindicated with FazaClo
* Patients who have been taking FazaCLo within the last three months
* Patients unable to comply with the required WBC/ANC monitoring schedule
* Patients unable to follow the physician's instructions
* Patients unable or unwilling to provide Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolled population consists of male and female patients with treatment-resistant schizophrenia of 18 years of age or older, already taking Clozaril (clozapine) or generic clozapine, or patients with treatment-resistant schizophrenia who have failed on other atypical antipsychotic drugs.
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Clinical changes in body weight in patients with treatment-resistant schizophrenia after initiating treatment with FazaClo
Clinical changes in salivation in patients with treatment-resistant schizophrenia after initiating treatment with FazaClo

SECONDARY OUTCOMES:
Changes in Clinical Global Impression (CGI) scale when compared to baseline

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pacific Neuropsychiatric Specialists, Costa Mesa, California
  - Gihwala & Associates, Gastonia, North Carolina